CLINICAL TRIAL: NCT04990908
Title: Systematic Screening for Primary Immunodeficiencies in Patients Admitted for Severe Infection in Pediatric Intensive Care Unit
Acronym: SPYSI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0378
Record Dates: First submitted 2021-07-05; First posted 2021-08-05 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-07

CONDITIONS: Severe Infection; Severe Immune Deficiency
Keywords: genetics; screening
MeSH Terms: conditions — Infections; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe infections in pediatric intensive care unit are not uncommon. Historically, the diagnosis of hereditary (primary) immune deficiency required a combination of recurrent clinical signs and biological stigmas. This paradigm is currently being questioned, and grows the hypothesis of a potential underlying genetic susceptibility in any severe infection. To date, the proportion of severe infections explained by an underlying immune deficiency is unknown.

The aim of this prospective study is to assess the incidence of primary immune deficiencies in children with severe infection, regardless of their etiology.

ELIGIBILITY:
Inclusion criteria:

* Inclusion age less than 16 years
* Inclusion age > 3 months of actual age for term infants and > 3 months for former preterm infants.
* Documented severe infection (bacterial, viral, fungal) at the University Hospital Center of Montpellier, Toulouse or Marseille
* Severe infections concerned by the study: any infection requiring hospitalization in pediatric intensive care (more than 24 hours) including:
* meninges or brain lesions, pleuro-pneumopathy, any infection associated with sepsis and/or an opportunistic germ, septic shock, etc.
* Encephalitis and encephalomyelitis of infectious origin
* Child benefiting from a social security system
* Collection of parental/legal representative consent

Exclusion criteria:

* Undocumented severe infections
* Acute bronchiolitis
* Children admitted with isolated SRV bronchiolitis without further complications from the infection;
* Previous comorbidity explaining the infection and/or stay in ICU/Continuing Care: Primary or known secondary immune deficiency; burns; risk factors for non-infectious epilepsy (encephalopathy, known epilepsy, head trauma), pneumonia caused by swallowing disorders or tracheotomy or chronic lung disease, asthma, meningitis favored by cochlear implants, breach of blood-brain barrier or neuromeningetic material, deep infection on implanted material or within 48h after surgery, cardiovascular decompensation; any other chronic conditions that may contribute to infection;
* Inability to obtain consent from parents/legal guardians.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
number of patients with primary immunodeficiency revealed after a severe infection in pediatric ICU or in neuropediatric unit | 1 day
  number of patients with primary immunodeficiency revealed after a severe infection in pediatric ICU or in neuropediatric unit

SECONDARY OUTCOMES:
Rate of to evaluate the sensitivity of our systematic screening | 1 day
  To evaluate the sensitivity of our systematic screening in relation to an approach scrupulously following the indications of other published studies for the screening of primary immunodeficiencies

OTHER OUTCOMES:
The number of immune deficiencies that have no other call point based on the list of warning signs of the Reference Center for Hereditary Immune Deficiencies (CEREDIH) | 1 day
  The number of immune deficiencies that have no other call point based on the list of warning signs of the Reference Center for Hereditary Immune Deficiencies (CEREDIH)

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC